CLINICAL TRIAL: NCT02625064
Title: Discovery of New Early Detection Biomarkers of Acute Respiratory Distress Syndrome
Acronym: ARDS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 20151030
Record Dates: First submitted 2015-11-24; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; biomarkers; proteomic
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: patient at High risk for ARDSp: Severe pneumonia and（PaO2/FIO2）>300mmHg
  Interventions: Other: Blood samples collection before treatment; Other: Blood samples collection after treatment; Other: laboratory biomarker proteomic analysis
- 2: patient at High risk for ARDSexp: Severe sepsis and without ARDS
  Interventions: Other: Blood samples collection before treatment; Other: Blood samples collection after treatment; Other: laboratory biomarker proteomic analysis
- 3: mild ARDS: PaO2/FiO2=201～300 mmHg，and PEEP or CPAP≤5 cm
  Interventions: Other: Blood samples collection before treatment; Other: Blood samples collection after treatment; Other: laboratory biomarker proteomic analysis
- 4: moderate ARDS: PaO2/FIO2=101～200 mmHg，且PEEP≥5 cm H2O
  Interventions: Other: Blood samples collection before treatment; Other: Blood samples collection after treatment; Other: laboratory biomarker proteomic analysis
- 5: severe ARDS: PaO2/FIO2≤100 mmHg，且PEEP≥10 cm H2O
  Interventions: Other: Blood samples collection before treatment; Other: Blood samples collection after treatment; Other: laboratory biomarker proteomic analysis

INTERVENTIONS:
Other: Blood samples collection before treatment
Other: Blood samples collection after treatment
Other: laboratory biomarker proteomic analysis

SUMMARY:
The goal of this project is to find a series novel biomarkers by differential proteomic techniques that can improve the early diagnosis and develop a more efficient therapy to enhance ARDS patient survival rate.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome(ARDS) has a very poor prognosis and high mortality. To improve the early diagnosis of ARDS, there is an urgent need for novel biomarkers of ARDS. The goal of this project is to find a series novel biomarkers by differential proteomic techniques that can improve the early diagnosis and develop a more efficient therapy to enhance ARDS patient survival rate. Clinical data and blood sample were recorded before treatment and after treatment. Acute Physiology And Chronic Health Evaluation III (APACHE III) scores were calculated at enrolment. Studying blood specimens from different period ARDS patients by proteomic analysis. It can provide information on a complex composition of proteins that are differentially expressed, which could be used for discovering high sensitivity and specificity ARDS biomarker.

ELIGIBILITY:
Inclusion Criteria:

* The Berlin definition of acute respiratory distress syndrome
* ATS definition of severe pneumonia

Exclusion Criteria:

* age below 18 years
* pregnancy
* Expected survival under 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at High risk for Extra-pulmonary ARDS and pulmonary ARDS; patients who have ARDS
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of serum proteins directly by proteomics analysis to identify new biomarkers of ARDS | baseline
Analysis of serum proteins directly by proteomics analysis to identify new biomarkers of ARDS | 1 month

SECONDARY OUTCOMES:
APACHE III score | baseline, 1week, 2 weeks
PaO2/FiO2 ratio | baseline, day 3, day 5, 1week, 2 weeks
Mortality or multi-organ failure | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pinhua Pan, MD, Doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Janz DR, Ware LB. Biomarkers of ALI/ARDS: pathogenesis, discovery, and relevance to clinical trials. Semin Respir Crit Care Med. 2013 Aug;34(4):537-48. doi: 10.1055/s-0033-1351124. Epub 2013 Aug 11. PMID 23934723
- [Background] Ware LB, Calfee CS. Biomarkers of ARDS: what's new? Intensive Care Med. 2016 May;42(5):797-799. doi: 10.1007/s00134-015-3973-0. Epub 2015 Jul 15. No abstract available. PMID 26174184
- [Background] Ware LB, Koyama T, Billheimer DD, Wu W, Bernard GR, Thompson BT, Brower RG, Standiford TJ, Martin TR, Matthay MA; NHLBI ARDS Clinical Trials Network. Prognostic and pathogenetic value of combining clinical and biochemical indices in patients with acute lung injury. Chest. 2010 Feb;137(2):288-96. doi: 10.1378/chest.09-1484. Epub 2009 Oct 26. PMID 19858233